CLINICAL TRIAL: NCT00284089
Title: Open-label Multicenter, Phase I/II Study Assessing the Safety and Efficacy of Ranibizumab (RFB002) in Japanese Patients With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD)
Brief Title: Safety and Efficacy of Ranibizumab in Japanese Patients With Subfoveal Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002A1201
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Subfoveal Choroidal Neovascularization(CNV) Secondary to Age-related Macular Degeneration (AMD)
Keywords: Subfoveal CNV, AMD, ranibizumab
MeSH Terms: interventions — Ranibizumab

ARMS (4):
- Group A: Ranibizumab 0.3 mg (Experimental): In the single dose phase, all patients randomized in Group A received a single intravitreal injection of 0.3 mg of ranibizumab into the study eye. Those patients who successfully completed this phase entered the multiple dose phase, where they received an intravitreal injection of 0.3 mg of ranibizumab once a month for an additional 11 months. Subsequently patients enrolling in the extension phase received an intravitreal injection of 0.3 mg of ranibizumab according to an individualized flexible interval regimen guided by monthly best corrected visual acuity scores and other ophthalmic examinations. In the extension phase patients received the same dose level as they received in the multiple dose phase of the study, for an average of 1.70 years.
  Interventions: Drug: Ranibizumab
- Group A: Ranibizumab 0.5 mg (Experimental): In the single dose phase, all patients randomized in Group A received a single intravitreal injection of 0.5 mg of ranibizumab into the study eye. Those patients who successfully completed this phase entered the multiple dose phase, where they received an intravitreal injection of 0.5 mg of ranibizumab once a month for an additional 11 months. Subsequently Group A patients enrolling in the extension phase received an intravitreal injection of 0.5 mg of ranibizumab according to an individualized flexible interval regimen guided by monthly best corrected visual acuity scores and other ophthalmic examinations. In the extension phase patients received the same dose level as they received in the multiple dose phase of the study, for an average of 1.93 years.
  Interventions: Drug: Ranibizumab
- Group B: Ranibizumab 0.3 mg (Experimental): Group B patients received a total of 12 monthly intravitreal injections of 0.3 mg of ranibizumab into the study eye in the multiple dose phase of the study. Group B patients who enrolled in the extension phase received an intravitreal injection of 0.3 mg of ranibizumab according to an individualized flexible interval regimen guided by monthly best corrected visual acuity scores and other ophthalmic examinations. In the extension phase patients received the same dose level as they received in the multiple dose phase of the study, for an average of 1.45 years.
  Interventions: Drug: Ranibizumab
- Group B: Ranibizumab 0.5 mg (Experimental): Group B patients received a total of 12 monthly intravitreal injections of 0.5 mg of ranibizumab into the study eye in the multiple dose phase of the study. Group B patients who enrolled in the extension phase received an intravitreal injection of 0.5 mg of ranibizumab according to an individualized flexible interval regimen guided by monthly best corrected visual acuity scores and other ophthalmic examinations. In the extension phase patients received the same dose level as they received in the multiple dose phase of the study, for an average of 1.36 years.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab was administered by intravitreal injection in the study eye. Intravitreal injection was performed by the investigator following slitlamp examination.
  Other Names: Lucentis

SUMMARY:
Open-label Multicenter, Phase I/II Study comprising three phases (single dose, multiple dose and extension phase), Assessing the Safety and Efficacy of Ranibizumab (RFB002) in Japanese Patients With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
The safety and tolerability of single intravitreal injections of ranibizumab was evaluated in patients enrolled in the single dose phase (Group A). Patients who successfully completed the single dose phase (i.e. did not experience a grade-3 targeted adverse event) could enter the multiple dose phase and receive ranibizumab injections for an additional 11 months. Simultaneously, the multiple dose phase was initiated in two parallel dose groups of additional patients (Group B), who received ranibizumab injections for 12 months. After patients in Group A and Group B had completed the multiple dose phase, all patients who provided written consent and were considered eligible based on the inclusion and exclusion criteria of the extension phase had the opportunity to continue on study treatment with the individualized flexible treatment regimen guided by monthly acuity scores and other ophthalmic examinations until approval of ranibizumab in Japan.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients 50 years of age or greater
2. Patients with primary or recurrent subfoveal CNV secondary to AMD
3. Patients who have a BCVA score between 73 and 24 letters in the study eye using ETDRS-like grading charts (approximately 20/40 to 20/320)

Exclusion Criteria

1. No prior treatment in the study eye with verteporfin, external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, or transpupillary thermotherapy

Extension Phase

Inclusion criteria:

1. Personally provided written informed consent to participate in the extension phase.
2. Patients with subfoveal CNV secondary to AMD who had completed the multiple dose phase in either of the ranibizumab groups (Group A or B).
3. Patients could participate in the extension phase even if they failed to do so on the day of the exit visit in the multiple dose phase (Group A and B), regardless of the time elapsed until the participation in the extension phase.

Exclusion criteria:

1. Received anti-angiogenic drugs (bevacizumab, pegaptanib, ranibizumab, anecortave acetate, corticosteroids or protein kinase C inhibitors, etc.) or
2. Participated in any clinical study of an investigational drug other than this one during the period between the exit visit of the multiple dose phase and the start in the extension phase, if they failed to be enrolled into the extension on the day of the exit visit. Patients were to be excluded even when the fellow eye was treated with any of these drugs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — Novartis
Locations (1):
- Novartis, Tokyo, Japan

REFERENCES:
- [Result] Tano Y, Ohji M; EXTEND-I Study Group. EXTEND-I: safety and efficacy of ranibizumab in Japanese patients with subfoveal choroidal neovascularization secondary to age-related macular degeneration. Acta Ophthalmol. 2010 May;88(3):309-16. doi: 10.1111/j.1755-3768.2009.01843.x. Epub 2010 Feb 16. PMID 20163368
- [Result] Tano Y, Ohji M; EXTEND-I Study Group. Long-term efficacy and safety of ranibizumab administered pro re nata in Japanese patients with neovascular age-related macular degeneration in the EXTEND-I study. Acta Ophthalmol. 2011 May;89(3):208-17. doi: 10.1111/j.1755-3768.2010.02065.x. Epub 2011 Jan 14. PMID 21232078

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 88 patients were enrolled in the study, 12 in Group A and 76 in Group B. The single dose phase of the study (Group A patients only) was completed prior to initiation of the multiple dose phase (Groups A and B).
Period: Single Dose Phase
Arm/Group | Group A: Ranibizumab 0.3 mg | Group A: Ranibizumab 0.5 mg | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Started | 6 | 6 | 0 (Group B patients did not participate in the Single Dose Phase of the study.) | 0 (Group B patients did not participate in the Single Dose Phase of the study.)
Completed | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Multiple Dose Phase
Arm/Group | Group A: Ranibizumab 0.3 mg | Group A: Ranibizumab 0.5 mg | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Started | 5 (1 subject chose to receive other treatment & discontinued before starting the multiple dose phase.) | 6 | 35 | 41
Completed | 4 | 6 | 31 | 37
Not Completed | 1 | 0 | 4 | 4
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 1 | 1
Period: Extension Phase
Arm/Group | Group A: Ranibizumab 0.3 mg | Group A: Ranibizumab 0.5 mg | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Started | 3 (Patients providing written consent & satisfying eligibility criteria could enter the extension phase) | 6 (Patients providing written consent & satisfying eligibility criteria could enter the extension phase) | 28 (Patients providing written consent & satisfying eligibility criteria could enter the extension phase) | 33 (Patients providing written consent & satisfying eligibility criteria could enter the extension phase)
Completed | 1 | 6 | 22 | 21
Not Completed | 2 | 0 | 6 | 12
Not completed — Adverse Event | 0 | 0 | 2 | 2
Not completed — condition no longer requires study drug | 2 | 0 | 2 | 7
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group B: Ranibizumab 0.3 mg: Group B patients received a total of 12 monthly intravitreal injections of 0.3 mg of ranibizumab into the study eye in the multiple dose phase of the study. Group B patients enrolled in the extension phase received an intravitreal injection of 0.3 mg of ranibizumab according to an individualized flexible interval regimen guided by monthly best corrected visual acuity scores and other ophthalmic examinations. In the extension phase patients received the same dose level as they received in the multiple dose phase of the study, for an average of 1.45 years.
- Total: Total of all reporting groups
Arm/Group | Group A: Ranibizumab 0.3 mg | Group A: Ranibizumab 0.5 mg | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg | Total
Number analyzed (Participants) | 6 | 6 | 35 | 41 | 88
Age, Customized [Number; unit: Participants] — Age demographics for those subjects enrolled in the single and multiple dose phases of the study.
  Participants
    50 to <65 years | 2 | 0 | 8 | 10 | 20
    65 to <75 years | 2 | 4 | 16 | 13 | 35
    75 to <85 years | 2 | 2 | 10 | 15 | 29
    >= 85 years | 0 | 0 | 1 | 3 | 4
Age, Customized [Number; unit: Participants] — Age demographics for those subjects enrolled in the extension phase of the study.
  Participants
    50 to <65 years | 1 | 0 | 7 | 10 | 18
    65 to <75 years | 1 | 4 | 14 | 10 | 29
    75 to <85 years | 1 | 2 | 6 | 12 | 21
    >= 85 years | 0 | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Gender demographics for those subjects enrolled in the single and multiple dose phases of the study.
  Participants
    Female | 1 | 1 | 9 | 8 | 19
    Male | 5 | 5 | 26 | 33 | 69
Gender [Number; unit: participants] — Gender demographics for those subjects enrolled in the extension phase of the study.
  participants
    Female | 0 | 1 | 9 | 5 | 15
    Male | 3 | 5 | 19 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Best Corrected Visual Acuity Score of the Study Eye at Month 6 in Group B
Description: The efficacy assessment was based on Group B patients. Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 2 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a starting test distance of 2 meters. The BCVA score is the number of letters read correctly by the patient, hence an increase in score indicates improvement in acuity.
Time Frame: Baseline and Month 6
Population: Intent-to treat (ITT) population for Group B patients consisted of all patients randomized in Group B that received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. The Last Observation Carried Forward (LOCF) was used to impute missing data at month 6 in the ITT analysis.
Measure: Mean (Standard Deviation); unit: Number of Letters
Groups:
- Group B: Ranibizumab 0.3 mg: Group B patients received a total of 12 monthly intravitreal injections of 0.3 mg of ranibizumab into the study eye in the multiple dose phase of the study.
- Group B: Ranibizumab 0.5 mg: Group B patients received a total of 12 monthly intravitreal injections of 0.5 mg of ranibizumab into the study eye in the multiple dose phase of the study.
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 35 | 41
Number of Letters
  Baseline | 47.6 (11.82) | 48.1 (10.75)
  Month 6 | 55.7 (13.16) | 57.1 (14.99)
  Change from Baseline | 8.1 (12.65) | 9.0 (9.62)

2. Secondary Outcome: Mean Change From Baseline in the Best Corrected Visual Acuity Score of the Study Eye at Month 12 in Group B
Description: The efficacy assessment was based on Group B patients. BCVA was assessed during all study visits using best correction determined from protocol refraction and ETDRS-like visual acuity testing charts at a starting test distance of 2 meters. The BCVA score is the number of letters read correctly by the patient, hence an increase in score indicates improvement in acuity.
Time Frame: Baseline and Month 12
Population: Intent-to treat (ITT) population for Group B patients consisted of all patients randomized in Group B that received at least one dose of study drug and had at least one post-baseline assessment of the efficacy variable. The Last Observation carried Forward (LOCF) was used to impute missing data at month 12 in the ITT analysis.
Measure: Mean (Standard Deviation); unit: Number of Letters
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 35 | 41
Number of Letters
  Baseline | 47.6 (11.82) | 48.1 (10.75)
  Month 12 | 57.1 (12.91) | 58.6 (15.44)
  Change from Baseline | 9.5 (12.79) | 10.5 (11.14)

3. Secondary Outcome: Categorical Analysis of Best Corrected Visual Acuity of the Study Eye at Month 6 and Month 12 in Group B
Description: BCVA measurements were taken in a sitting position using best correction determined from protocol refraction and ETDRS-like visual acuity testing charts at a starting test distance of 2 meters.
Time Frame: Baseline, Month 6 and Month 12
Population: ITT population, using LOCF.
Measure: Number; unit: Participants
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 35 | 41
Participants
  Loss of < 15 letters from Baseline at month 6 | 34 | 41
  Loss of < 15 letters from Baseline at month 12 | 34 | 41
  Gain of ≥15 letters from Baseline at month 6 | 12 | 10
  Gain of ≥15 letters from Baseline at month 12 | 13 | 13
  Loss of ≥30 letters from Baseline at month 6 | 0 | 0
  Loss of ≥30 letters from Baseline at month 12 | 0 | 0
  Visual acuity < 34 letters at Month 6 | 2 | 2
  Visual acuity < 34 letters at Month 12 | 2 | 1

4. Secondary Outcome: Extension Phase: Mean Change From Month 12 (Start of Extension Phase) in Best Corrected Visual Acuity Score of the Study Eye at Last Visit of Extension Phase in Group B.
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 2 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a starting test distance of 2 meters. The BCVA score is the number of letters read correctly by the patient, hence an increase in score indicates improvement in acuity.
Time Frame: Month 12 (start of extension phase) and last visit of extension phase. Duration in the extension phase varied depending on the study entry. The mean duration of treatment was 1.45 years in the 0.3 mg group and 1.36 years in the 0.5 mg dose group.
Population: The analysis population included all enrolled patients in the extension phase. For the analysis of the results of the extension phase, all data are presented as observed. Patients must have values both at Month 12 and Last Visit to be included.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 28 | 33
Letters
  Baseline | 47.9 (12.59) | 50.0 (10.38)
  Month 12 | 59.1 (11.69) | 59.8 (15.07)
  Last visit | 55.4 (17.14) | 57.6 (15.36)
  Change from Month 12 | -3.6 (14.82) | -2.2 (7.92)

5. Secondary Outcome: Extension Phase: Categorical Analysis of Best Corrected Visual Acuity of the Study Eye at Last Visit of Extension Phase in Group B
Description: BCVA measurements were taken in a sitting position using best correction determined from protocol refraction and ETDRS-like visual acuity testing charts at a starting test distance of 2 meters. The following categories were evaluated:
  * Participants with a BCVA score loss of fewer than 15 letters from baseline at Last Visit
  * Participants with a BCVA score loss of 30 or more letters from baseline at Last Visit
  * Participants with a BCVA score gain of 15 or more letters from baseline at Last Visit
  * Participants with a BCVA score of less than 34 letters at Last Visit
Time Frame: Baseline and last visit of extension phase - Duration in the extension phase varied depending on the study entry. The mean duration of treatment was 1.45 years in the 0.3 mg group and 1.36 years in the 0.5 mg dose group.
Population: Includes patients enrolled in the extension phase, observed data.
Measure: Number; unit: Participants
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 28 | 33
Participants
  Loss of < 15 letters from Baseline | 24 | 32
  Gain of ≥15 letters from Baseline | 9 | 9
  Loss of ≥30 letters from Baseline | 1 | 1
  Visual acuity < 34 letters | 3 | 1

6. Secondary Outcome: Mean Change From Baseline in Total Area of Choroidal Neovascularization of the Study Eye in Group B
Description: Choroidal Neovascularization was assessed by fluorescein angiography in conjunction with color fundus photography. Analysis was performed by the central reading center. The area of Choroidal Neovascularization is expressed as Macular Photocoagulation Study standard Disc Areas (DA; equivalent to 2.54 mm^2 on the retina).
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: Intent-to treat (ITT) population for Group B patients consisted of all patients randomized in Group B that received at least one dose of study drug and had at least one post-baseline assessment. The Last Observation Carried Forward (LOCF) was used to impute missing data.
Measure: Mean (Standard Deviation); unit: disc areas
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 35 | 41
disc areas
  Baseline [N=35, 41] | 2.11 (1.10) | 2.03 (1.66)
  Mean change from Baseline at Month 3 [N=34, 40] | -0.10 (0.95) | 0.13 (0.75)
  Mean change from Baseline at Month 6 [N=34, 40] | -0.15 (0.97) | 0.04 (0.76)
  Mean change from Baseline at Month 9 [N=34, 40] | -0.23 (0.97) | 0.21 (0.90)
  Mean change from Baseline at Month 12 [N=34, 40] | -0.16 (1.01) | 0.23 (1.08)

7. Secondary Outcome: Mean Change From Baseline in Total Area of Leakage From CNV Plus Staining of Retinal Pigment Epithelium of the Study Eye in Group B
Description: Area of leakage from CNV plus staining of retinal pigment epithelium was assessed by fluorescein angiography in conjunction with color fundus photography. Analysis was performed by the central reading center. The total area is expressed as Macular Photocoagulation Study standard Disc Areas (DA; equivalent to 2.54 mm^2 on the retina).
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: disc areas
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 35 | 41
disc areas
  Baseline [N=35, 41] | 2.31 (1.17) | 2.49 (1.54)
  Mean change from Baseline at Month 3 [N=34, 40] | -0.76 (0.85) | -0.74 (1.21)
  Mean change from Baseline at Month 6 [N=34, 40] | -1.21 (0.87) | -1.10 (1.19)
  Mean change from Baseline at Month 9 [N=34, 40] | -1.39 (1.02) | -1.26 (1.45)
  Mean change from Baseline at Month 12 [N=34, 40] | -1.50 (1.08) | -1.39 (1.48)

8. Secondary Outcome: Percentage of Participants in Group B With Absence of Leakage in the Study Eye at Month 3, 6, 9 and 12.
Description: Area of leakage was assessed by fluorescein angiography in conjunction with color fundus photography. Analysis was performed at the central reading center.
Time Frame: Months 3, 6, 9 and 12
Population: Intent-to treat (ITT) population for Group B patients consisted of all patients randomized in Group B that received at least one dose of study drug and for whom data was available. The Last Observation Carried Forward (LOCF) was used to impute missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 34 | 40
Percentage of participants
  Month 3 | 2.9 | 7.5
  Month 6 | 8.8 | 15.0
  Month 9 | 26.5 | 25.0
  Month 12 | 35.3 | 35.0

9. Secondary Outcome: Mean Change From Baseline in Foveal Retinal Thickness of the Study Eye in Group B
Description: Foveal retinal thickness was assessed by Optical Coherence Tomography (OCT) at a subset of the study sites and was analyzed by the central reading center.
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: The analysis includes Group B Intent-to treat (ITT) population, observed data. OCT was performed in a total of 58 patients at selected sites.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 28 | 30
micrometers
  Baseline [N=28, 30] | 336.7 (195.3) | 370.7 (171.9)
  Mean change from Baseline at Month 3 [N=27, 29] | -124.4 (141.6) | -195.6 (187.5)
  Mean change from Baseline at Month 6 [N=26, 28] | -142.9 (199.3) | -225.6 (192.2)
  Mean change from Baseline at Month 9 [N=26, 27] | -188.4 (190.1) | -245.4 (203.1)
  Mean change from Baseline at Month 12 [N=26, 26] | -194.0 (199.8) | -257.8 (209.8)

10. Secondary Outcome: Mean Change From Baseline in Total Retinal Volume of the Study Eye in Group B
Description: Total retinal volume was assessed by Optical Coherence tomography (OCT) at a subset of the study sites and was analyzed by the central reading center.
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: OCT was performed in a total of 58 patients at selected sites. Group B Intent-to treat (ITT) population, observed data only are included. The assessed sample size was small for total retinal volume data because the central reading center judged "Can not grade" due to retinal pigment epithelium disruption associated with CNV secondary to AMD.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group B: Ranibizumab 0.3 mg | Group B: Ranibizumab 0.5 mg
Number analyzed (Participants) | 28 | 30
micrometers
  Baseline [N=11, 11] | 7.23 (0.84) | 7.36 (0.97)
  Mean change from Baseline at Month 3 [N=7, 7] | -0.78 (0.74) | -0.67 (0.71)
  Mean change from Baseline at Month 6 [N=6, 6] | -0.52 (0.60) | -0.92 (0.96)
  Mean change from Baseline at Month 9 [N=4, 5] | -0.48 (0.03) | -0.28 (0.83)
  Mean change from Baseline at Month 12 [N=6, 6] | -0.95 (1.14) | -0.42 (0.67)

ADVERSE EVENTS:
Time Frame: The timeframe for the Core Phase (Single and Multiple Dose Phases) was 12 months. For the Extension Phase adverse event data was collected from Month 12 through to the Last Visit (the maximum time on study was 35 months total).
Groups:
- Core Group A+B: Ranibizumab 0.3 mg: "Core" means Single and Multiple Dose Phases. Group A patients received a single intravitreal injection of 0.3 mg of ranibizumab into the study eye, followed by 11 additional intravitreal injections of 0.3 mg of ranibizumab once a month. Group B patients received a total of 12 monthly intravitreal injections of 0.3 mg of ranibizumab into the study eye.
- Core Group A+B: Ranibizumab 0.5 mg: "Core" means Single and Multiple Dose Phases. Group A patients received a single intravitreal injection of 0.5 mg of ranibizumab into the study eye, followed by 11 additional intravitreal injections of 0.5 mg of ranibizumab once a month. Group B patients received a total of 12 monthly intravitreal injections of 0.5 mg of ranibizumab into the study eye.
- Extension Group A+B: Ranibizumab 0.3 mg: In the extension phase, enrolled patients received an intravitreal injection of 0.3 mg ranibizumab according to an individualized flexible interval regimen guided by monthly best corrected visual acuity scores and other ophthalmic examinations. In the extension phase patients received the same dose level as they received in the multiple dose phase of the study, for an average of 1.45 years.
- Extension Group A+B: Ranibizumab 0.5 mg: In the extension phase, all patients received an intravitreal injection of 0.5 mg ranibizumab according to an individualized flexible interval regimen guided by monthly best corrected visual acuity scores and other ophthalmic examinations. In the extension phase patients received the same dose level as they received in the multiple dose phase of the study, for an average of 1.36 years.
Arm/Group | Core Group A+B: Ranibizumab 0.3 mg | Core Group A+B: Ranibizumab 0.5 mg | Extension Group A+B: Ranibizumab 0.3 mg | Extension Group A+B: Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 5/41 | 8/47 | 5/31 | 8/39
Other Adverse Events (participants affected / at risk) | 38/41 | 43/47 | 27/31 | 28/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Group A+B: Ranibizumab 0.3 mg (N=41) | Core Group A+B: Ranibizumab 0.5 mg (N=47) | Extension Group A+B: Ranibizumab 0.3 mg (N=31) | Extension Group A+B: Ranibizumab 0.5 mg (N=39)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Cataract (Fellow eye) (Eye disorders) | 1 | 1 | 0 | 0
Corneal oedema (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Eye pain (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Glaucomatocyclitic crises (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Macular degeneration (Fellow eye) (Eye disorders) | 1 | 0 | 0 | 0
Macular degeneration (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Retinal detachment (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Fellow eye) (Eye disorders) | 0 | 0 | 0 | 1
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced transiently (Study eye) (Eye disorders) | 0 | 2 | 0 | 0
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocele (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 1
Overdose (Study eye) (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Intraocular pressure increased (Study eye) (Investigations) | 0 | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Group A+B: Ranibizumab 0.3 mg (N=41) | Core Group A+B: Ranibizumab 0.5 mg (N=47) | Extension Group A+B: Ranibizumab 0.3 mg (N=31) | Extension Group A+B: Ranibizumab 0.5 mg (N=39)
Conjunctival haemorrhage (Study eye) (Eye disorders) | 30 | 28 | 13 | 14
Conjunctival hyperaemia (Study eye) (Eye disorders) | 8 | 8 | 2 | 1
Conjunctivitis allergic (Fellow eye) (Eye disorders) | 0 | 0 | 0 | 2
Conjunctivitis allergic (Study eye) (Eye disorders) | 1 | 1 | 0 | 2
Eye pain (Study eye) (Eye disorders) | 9 | 10 | 2 | 0
Myodesopsia (Study eye) (Eye disorders) | 0 | 0 | 0 | 3
Ocular hyperaemia (Study eye) (Eye disorders) | 0 | 3 | 0 | 0
Polypoidal choroidal vasculopathy (Fellow eye) (Eye disorders) | 0 | 0 | 2 | 0
Punctate keratitis (Study eye) (Eye disorders) | 7 | 4 | 1 | 1
Retinal detachment (Study eye) (Eye disorders) | 5 | 2 | 2 | 5
Retinal haemorrhage (Fellow eye) (Eye disorders) | 3 | 5 | 6 | 2
Retinal haemorrhage (Study eye) (Eye disorders) | 12 | 5 | 9 | 10
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 3 | 1 | 0
Vitreous detachment (Study eye) (Eye disorders) | 3 | 0 | 0 | 0
Vitreous floaters (Study eye) (Eye disorders) | 1 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 1 | 1 | 1
Dental caries (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 7 | 10 | 6 | 9
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Intraocular pressure increased (Study eye) (Investigations) | 2 | 6 | 2 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0
Headache (Nervous system disorders) | 4 | 1 | 2 | 1
Prostatomegaly (Reproductive system and breast disorders) | 3 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0
Hypertension (Vascular disorders) | 3 | 1 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.